CLINICAL TRIAL: NCT06384222
Title: Hyperpolarized (HP) 13C Pyruvate Magnetic Resonance Imaging (MRI) as a Response Monitoring Tool in Patients With High-Risk Prostate Cancer Receiving Neoadjuvant Therapy
Brief Title: Hyperpolarized (HP) 13C Pyruvate Magnetic Resonance Imaging (MRI) for Response Monitoring to Neoadjuvant Abiraterone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ivan de Kouchkovsky, MD (Other)
Responsible Party: Sponsor-Investigator, Ivan de Kouchkovsky, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 235513; NCI-2024-03418 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: High Risk Prostate Carcinoma; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; abiraterone; Prednisone; Pyruvic Acid; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Abiraterone/Prednisone, Hyperpolarized (HP) 13C Pyruvate) (Experimental): Neoadjuvant abiraterone (1000mg) will be administered for three 28-day cycles, in conjunction with 5mg of prednisone. Participants will undergo a paired multi-parametric/hyperpolarized MRI of the prostate at screening, cycle 2 day 1, and after completion of neoadjuvant therapy. With each scan, a hyperpolarized 13C-pyruvate injection will be administered and an endorectal coil will be inserted prior to and removed after completion of the 1H and 13C MR exam using standard institutional procedures for preparation and placement for enhanced imaging. A planned, non-investigational RP will be completed within 7-56 days after last dose/discontinuation of neoadjuvant study drug. Participants will be followed up until death, withdrawal of consent, or end of study, whichever occurs first.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Hyperpolarized [1-13C] pyruvate (HP 13C); Procedure: Magnetic Resonance Imaging (MRI); Procedure: Non-investigational radical prostatectomy (RP); Procedure: Prostate-Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) PET/Computerized tomography (CT)

INTERVENTIONS:
Drug: Abiraterone acetate — Given orally
  Other Names: Abiraterone
Drug: Prednisone — Given orally
  Other Names: Rayos
Drug: Hyperpolarized [1-13C] pyruvate (HP 13C) — Given IV
  Other Names: Hyperpolarized 13C
Procedure: Magnetic Resonance Imaging (MRI) — Imaging procedure
  Other Names: MRI; MR
Procedure: Non-investigational radical prostatectomy (RP) — Planned, standard of care surgical procedure occurring outside of this study.
  Other Names: Radical prostatectomy
Procedure: Prostate-Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) PET/Computerized tomography (CT) — Imaging procedure

SUMMARY:
This study will evaluate the use of hyperpolarized 13C MRI (HP 13C MRI) and the HP-derived 13C pyruvate-to-lactate conversion rate constant (kPL) as an early response biomarker in men with treatment-naïve, high-risk, localized or locally advanced prostate cancer receiving neoadjuvant therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate on-treatment changes in HP 13C MRI derived kPL as an early response biomarker in men with high-risk localized or locally advanced prostate cancer receiving neoadjuvant abiraterone/prednisone prior to radical prostatectomy (RP).

SECONDARY OBJECTIVES:

I. To evaluate the pathologic complete response/minimal residual disease rate at the time of radical prostatectomy following 12 weeks of neoadjuvant abiraterone/prednisone in patients with high-risk localized or locally advanced prostate cancer.

II. To determine the safety and tolerability of neoadjuvant abiraterone/prednisone in patients with high-risk localized or locally advanced prostate cancer planning to undergo radical prostatectomy (RP).

III. To assess time to biochemical recurrence following radical prostatectomy after 12 weeks of neoadjuvant abiraterone/prednisone IV. To assess prostate-specific antigen (PSA) response to neoadjuvant abiraterone/prednisone prior to RP.

EXPLORATORY OBJECTIVES:

I. To assess the diagnostic performances of multiparametric MRI (mpMRI) and hyperpolarized 13C MRI (HP13C MRI) for pathological response at the time of RP II. To investigate the association between early changes in intratumoral metabolism (HP 13C derived pyruvate-to-lactate conversion rate kPL) on neoadjuvant abiraterone with PSA nadir. III. To evaluate associations between baseline genomic and transcriptional features, changes in intratumoral kPL, and pathologic response at the time of radical prostatectomy.

OUTLINE:

Participants will receive 12 weeks of neoadjuvant abiraterone/prednisone. After completion of neoadjuvant therapy, participants will proceed to radical prostatectomy. Participants will be followed for up to 5 years every 3 months for the first year following RP, then every 6 months until death, biochemical recurrence or initiation of additional prostate cancer directed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age
2. Histologically confirmed adenocarcinoma of the prostate with archival biopsy tissue (collected within 12 months of cycle 1 day 1 of treatment) available for genomic profiling.

   a. Tumor tissue does not need to be retrieved but rather identified and available upon later request for future pathologic review and possible correlative studies.
3. High-risk disease defined as meeting 1 or more of the 3 following criteria:

   1. Gleason grade group >=4; or
   2. Pelvic node involvement by conventional imaging or PSMA PET imaging (cN1); or
   3. Tumor stage T3 or higher (i.e. tumor extension outside of the prostate, or spread to tissues near the prostate other than the seminal vesicles, such as the bladder or wall of the pelvis) as determined by conventional imaging (including prostate MRI), transrectal ultrasound or PSMA PET imaging.
4. No evidence of distant metastatic disease as determined by PSMA PET/CT or PET/MR. Nodal disease below the iliac bifurcation (clinical stage N1) is not an exclusion.
5. Participants must be planning to undergo radical prostatectomy (RP) with or without pelvic lymph node dissection and considered surgically resectable by urologic evaluation at the time of study entry. Adjuvant therapy following RP will be allowed per treating provider discretion.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Demonstrates adequate organ function as defined below:

   1. Absolute neutrophil count (ANC) >=1,500/microliter (mcL).
   2. Platelets >=100,000/mcL, independent of transfusions/growth factors within 3 months of treatment start.
   3. Total bilirubin within normal institutional limits, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits.
   4. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) <=3 X institutional upper limit of normal.
   5. Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <=3 X institutional upper limit of normal.
   6. Estimated creatinine clearance >=40 mL/min (by the Cockcroft Gault equation).
8. Ability to understand and the willingness to sign a written informed consent document.
9. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
10. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
11. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
12. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
13. Abiraterone may cause fetal harm when administered to a pregnant woman. The effects of hyperpolarized [1-13C]pyruvate on the developing human fetus are unknown. For this reason, men treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation and for 8 weeks after last administration of study treatment.

Exclusion Criteria:

1. Participants unwilling or unable to undergo MR imaging, including patients with contraindications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
2. Participants who cannot tolerate or have contra-indications to endorectal coil insertion; for example, patients with a prior abdominoperineal resection of the rectum or latex allergy. The use of an endorectal coil may be waived at the discretion of the Principal Investigator upon review of available imaging with radiology, in which case this exclusion criteria will not apply.
3. Participants with contra-indications to injection of gadolinium contrast; for example, participants with prior documented allergy or those with inadequate renal function.
4. Metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging.
5. Poorly controlled hypertension, with blood pressure at study entry >160 mmHg systolic or >100 mmHg diastolic.
6. Congestive heart failure with New York Heart Association (NYHA) status >=2.
7. A history of clinically significant EKG abnormalities, including QT prolongation, a family history of prolonged QT interval syndrome, or myocardial infarction within 6 months of study entry.
8. Has received prior prostate cancer therapy.

   a. Prior 5-alpha reductase inhibitors (e.g. finasteride, dutasteride) allowed if discontinued at least 3 weeks prior to first dose.
9. Is currently receiving any other investigational agent(s) or has participated in a study of an investigational product and received study treatment or used an investigational device within 2 weeks of the first dose of treatment.
10. Concurrent use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole,clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, indinavir, nelfinavir, voriconazole) or inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean changes in intratumoral pyruvate-to-lactate conversion rate constant (kPL) | Up to 4 weeks
  Mean changes in intratumoral kPL from baseline to 4 weeks will be reported. For participants with >1 intraprostatic lesions detected on baseline scan, change in kPL will be calculated on using the lesion with the highest initial kPL.

SECONDARY OUTCOMES:
Pathological response rate | Up to 3 months
  Pathological response rate is defined as the rate of combined pathological complete response (pCR) or minimal residual disease (MRD) at radical prostatectomy (RP). The point estimate and 95% confidence intervals will be reported. A pCR is defined as the absence of tumor on the gross specimen o MRD is defined as residual tumors with cross-sectional diameter of <=0.5cm.
Proportion of participants with treatment-related adverse events (TRAE) | Up to 3 months
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria. Proportion of participants reporting treatment-related adverse events will be reported.
Proportion of participants completing non-interventional radical prostatectomy (RP) | Up to 8 weeks following completion of neoadjuvant treatment.
  Proportion of patients successfully undergoing planned, non-interventional RP following neoadjuvant therapy will be reported.
Median Time to Biochemical Recurrence | Up to 5 years
  The Kaplan-Meier method will be used to estimate the median time to biochemical recurrence (along with 95% confidence intervals). Biochemical recurrence will be defined as a serum PSA >=0.2 ng/mL confirmed on two separate occasions (with time of biochemical recurrence defined as the date of the first serum PSA >=0.2 ng/mL). Participants deceased or initiated on a prostate cancer (PC)-directed therapy prior to biochemical recurrence will be censored at the time of death or initiation of PC-directed therapy. Similarly, participants removed from the trial prior to biochemical recurrence will be censored at the time of study removal.
Proportion of participants with a >=50% decline in PSA level from baseline (PSA50) response | Up to 4 months
  Proportion of patients with a PSA50 response defined as a >=50% decline in PSA level from baseline during neoadjuvant treatment will be reported.
Proportion of participants with a >=90% decline in PSA level from baseline (PSA90) response | Up to 4 months
  Proportion of patients with a PSA90 response defined as a >=90% decline in PSA level from baseline during neoadjuvant treatment will be reported.
Mean PSA nadir | Up to 4 months
  The mean PSA nadir for participants while on neoadjuvant therapy will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan de Kouchkovsky, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No